CLINICAL TRIAL: NCT02241954
Title: Ertical Expandable Prosthetic Titanium Rib (VEPTR) for Thoracic Insufficiency Syndrome
Brief Title: Vertical Expandable Prosthetic Titanium Rib (VEPTR) for Thoracic Insufficiency Syndrome
Acronym: VEPTR
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey Martus, Assistant Professor of Orthopaedics, Vanderbilt University Medical Center
Other Study IDs: 091371
Record Dates: First submitted 2014-09-03; First posted 2014-09-16 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Thoracic Insufficiency Syndrome (TIS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Expansion Thoracoplasty: The rib prosthesis is lengthened periodically to correct the concavity of the deformity, expanding the volume of the hypoplastic thorax and improving associated spinal deformity. This device has been FDA approved by a Humanitarian Device Exemption and is described as a Vertical Expandable Prosthetic Titanium Rib (VEPTR). An updated version of the VEPTR, the VEPTR II, may be used instead depending on the physician's preference and the patient's anatomy. The VEPTR II device has greater size range and modularity of implants than the original VEPTR.
  Interventions: Device: Synthes VEPTR (Vertical Expandable Prosthetic Titanium Rib)

INTERVENTIONS:
Device: Synthes VEPTR (Vertical Expandable Prosthetic Titanium Rib)

SUMMARY:
The hypothesis of the study is that individuals with poor pulmonary function secondary to TIS will benefit from expansion thoracoplasty. The investigators specific aims are to:

1. Record pulmonary function and thoracic volume of TIS patients at enrollment and with serial observation
2. Offer expansion thoracoplasty therapy to TIS patients with

   1. poor pulmonary function at enrollment
   2. progressive decline in pulmonary function
   3. progressive chest wall and/or spinal deformity
   4. lack of appropriate increase in thoracic volume during growth
3. Document efficacy of expansion thoracoplasty for TIS patients

DETAILED DESCRIPTION:
Study procedures

1. Patient Identification & Enrollment Patients meeting the inclusion criteria will be invited to enroll in the study as described above.
2. Serial clinical observation

   Patients will be followed over time for progression of thoracic insufficiency indicators:
   * Worsening respiratory status oFrequent respiratory infections oElevated resting respiratory rate oEase of fatigability oHypoxia and hypercapnia oMarionette sign (trunk and shoulder elevation and depression with respiration)
   * Primary diaphragmatic breathing (loss of chest wall mobility)
   * Progressive scoliosis
   * Failure of thoracic dimensions to increase with growth

   Patients with progressive thoracic insufficiency will be offered surgical intervention with expansion thoracoplasty utilizing the VEPTR device.

   Studies which are standard of care for TIS will be utilized to assess patients. Routine standard of care studies will be obtained:
   1. MRI of the spine will be obtained at presentation.
   2. Chest CT scan (every 2 years, or less frequently if clinically indicated)
   3. AP/Lat spine xrays (to include the chest wall)

   <!-- -->

   1. Will be obtained every 6 months - 12 months
   2. If a patient has a VEPTR implantation, the typical schedule of radiographs would include immediate postoperative xrays (the day of surgery and/or early postoperative period) and at 6 weeks, 12 weeks, and 6 months postoperative.
   3. VEPTR lengthening will typically take place every 6 months after the initial VEPTR implantation.

   i.Xrays will be obtained every 6 months in association with the VEPTR lengthening.

   ii.Once VEPTR lengthening is no longer clinically indicated, the patients will be followed with xrays every 6-24 months until skeletal maturity.

   d.Pulmonary function tests (spirometry) will be obtained every 6-12 months in children who are old enough to participate (typically > age 4 years).

   e.Arterial and/or capillary blood gases

   a.Blood gases will be obtained every 6-12 months if clinically indicated and perioperatively for VEPTR implantation / lengthening.

   f.Routine vital signs including resting pulse oximetry (SaO2)

   a.Will be assessed at clinic visits and perioperatively g.All of the above mentioned studies will be obtained more or less frequently as clinically indicated.
3. Expansion thoracoplasty with VEPTR implantation and subsequent lengthening with the VEPTR will be performed following informed consent. The surgical technique will be as described by Campbell.3 The VEPTR device will be lengthened at 6 to 12 month intervals until thoracic and spinal deformities have stabilized radiographically.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients, age range from 6 months - 17 years with thoracic insufficiency syndrome (TIS) will be considered for inclusion. Categories of TIS include:

  1. Flail chest syndrome
  2. Constrictive chest wall syndrome (rib fusions and scoliosis)
  3. Hypoplastic thorax syndrome (Jeune's syndrome, achondroplasia, Jarcho-levin syndrome, Ellis van Creveld syndrome)
  4. Progressive scoliosis/kyphosis of congenital, neurogenic, or idiopathic origin without rib anomaly
  5. Early onset scoliosis without rib anomaly at high risk for progression

Exclusion Criteria:

* Failure to meet inclusion criteria.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients, age range from 6 months to 17 years with thoracic insufficiency syndrome (TIS). Categories of TIS include:
  1. Flail chest syndrome
  2. Constrictive chest wall syndrome (rib fusions and scoliosis)
  3. Hypoplastic thorax syndrome (Jeune's syndrome, achondroplasia, Jarcho-levin syndrome, Ellis van Creveld syndrome)
  4. Progressive scoliosis/kyphosis of congenital, neurogenic, or idiopathic origin without rib anomaly
  5. Early onset scoliosis without rib anomaly at high risk for progression
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-11-11 (Actual); Primary Completion 2018-03-25 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Pulmonary function and thoracic volume of TIS patients | Enrollment (Baseline), Serial Observation Postop (Change from baseline at: 6 week, 12 week, 6 month, and every 6 months after that.)
  1)Record pulmonary function and thoracic volume of TIS patients at enrollment and with serial observation postoperatively (Change from baseline at: 6 week, 12 week, 6 month, and every 6 months after that.)
ffer expansion thoracoplasty therapy to TIS patients meeting certain criteria (provided in description below) | Enrollment (Baseline), Serial Observation Postop (Change from baseline at: 6 week, 12 week, 6 month, and every 6 months after that.)
  Offer expansion thoracoplasty therapy to TIS patients with
  * poor pulmonary function at enrollment
  * progressive decline in pulmonary function
  * progressive chest wall and/or spinal deformity
  * lack of appropriate increase in thoracic volume during growth
Document efficacy of expansion thoracoplasty for TIS patients | Enrollment (Baseline), Serial Observation Postop (Change from baseline at: 6 week, 12 week, 6 month, and every 6 months after that.)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Martus, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No